CLINICAL TRIAL: NCT01059058
Title: Treatment of White Spot Lesions After Orthodontic Treatment: A Practice-based Randomized Controlled Trial
Brief Title: Study of Treatments Used for White Spot Lesions After Orthodontic Treatment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Pacific NW Dental Practice-Based Research Network (Network)
Responsible Party: Principal Investigator, Greg Huang, Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 37062-E/B
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Tooth Demineralization
Keywords: MI Paste Plus; Fluoride Varnish; CPP-ACP; White Spot Lesions; Remineralization; Orthodontic Treatment
MeSH Terms: conditions — Tooth Demineralization | interventions — casein phosphopeptide-amorphous calcium phosphate nanocomplex; Home Care Services

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Test Group A: MI Paste Plus Group (Active Comparator)
  Interventions: Procedure: MI Paste Plus; Procedure: Normal Home Care
- Test Group B: Fluoride Varnish Group (Active Comparator)
  Interventions: Procedure: PreviDent Fluoride Varnish; Procedure: Normal Home Care
- Control Group (Placebo Comparator)
  Interventions: Procedure: Normal Home Care

INTERVENTIONS:
Procedure: MI Paste Plus — A trained staff member from the NW PRECEDENT dental/orthodontic office will give 3 tubes of MI Paste Plus (10% CPP-ACP + 900 ppm Fluoride paste) and instructions to the subject for home use. A pea-sized amount for each arch will be applied 2x/day for 8 weeks. Subjects will apply cream topically to the teeth with their finger or a cotton swab, spread around with their tongue, hold for 1-2 minutes, then expectorate.
  Other Names: CPP-ACP
  Arms: Test Group A: MI Paste Plus Group
Procedure: PreviDent Fluoride Varnish — A trained staff member from the NW PRECEDENT dental/orthodontic office will provide a SINGLE application of PreviDent fluoride varnish (22,600 ppm Fluoride) to the subject. The total dosage will be 0.5 mL.
  Other Names: Fluoride varnish
  Arms: Test Group B: Fluoride Varnish Group
Procedure: Normal Home Care — Subjects will receive non-prescription fluoride toothpaste (1100 ppm Fluoride) and oral hygiene instructions. The dosage will be 1/2 inch strip of paste 2x/day for 8 weeks. Subjects will apply paste to a toothbrush and brush teeth thoroughly for at least 1 minute then expectorate.
  Other Names: Home care

SUMMARY:
The purpose of this study is to learn more about the management of white spot lesions that occur after orthodontic treatment. White spot lesions generally improve slightly with time. To date, there is no proven method to help white spot lesions improve faster. Two treatments, called MI Paste Plus and fluoride varnish, have shown some potential benefits in a laboratory setting but have not undergone testing in a clinical setting. Approximately 240 subjects are to be enrolled in this study. The study will take place in approximately 30 dental and orthodontic offices across Idaho, Montana, Oregon, Utah, and Washington as part of Northwest PRECEDENT, a five-state research network that was created to study the practical issues facing dentists/orthodontists and their patients, and to provide information that will improve the quality of oral health care as a whole. Researchers at the University of Washington and Oregon Health & Science University share management and oversight of the network and research projects.

DETAILED DESCRIPTION:
White spot lesions (WSL), caused by the decalcification of enamel, are a common and unfortunate sequela of orthodontic treatment. If not addressed, WSL may progress to caries and frank cavitation of the enamel surface. Once formed, white spot lesions compromise esthetics and can be extremely difficult or even impossible to reverse. Many clinicians consider a high-dose fluoride application to be the first step in treatment of WSL in order to arrest areas of decalcification. However, some believe that while remineralization with high levels of fluoride may repair the surface of enamel, it may possibly block remineralization of the deeper areas of enamel. This, in turn, may hamper efforts to normalize the appearance of WSL.

Casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) containing products are a recently proposed therapy for the treatment of white spots following orthodontic treatment. CPP is thought to stabilize and localize calcium, fluoride, and phosphate at the tooth surface in a slow-release amorphous form, thus enhancing deeper remineralization of WSL. Products containing CPP-ACP are currently marketed under various names, including MI Paste Plus (which also contains fluoride). Few in vivo studies have investigated the effectiveness of various remineralization products to address WSL after orthodontics. This project is a single-blind, randomized clinical trial with three arms - MI Paste Plus for an 8-week duration, a single application of Duraphat Fluoride Varnish with reassessment at 8 weeks, and normal home care for an 8 week period. Subjects will be recruited at their regularly scheduled orthodontic appointments, with eligible subjects being up to 2 years post-removal of fixed orthodontic appliances.

This project is intended to answer four questions regarding the management of white spot lesions.

Specific Aim 1: to compare the effectiveness MI Paste Plus and Duraphat Fluoride Varnish to a standard oral hygiene/toothpaste regimen in improving the appearance of WSL after orthodontic treatment.

Specific Aim 2: to investigate subjects' self-assessment of improvement in each of the three arms.

Specific Aim 3: to investigate variables (such as age, gender, time since fixed orthodontic appliance removal, compliance, oral hygiene practices, etc) that may influence WSL improvement.

Specific Aim 4: to investigate the short-term changes in WSL from the day of orthodontic appliance removal until the day of retainer delivery (usually 2 - 7 days).

This study will provide valuable evidence on the management of WSL after orthodontic treatment. As previously stated, WSL lesions are quite common and difficult to reverse, so it is important to conduct rigorous clinical research in an effort to develop effective strategies.

This study will be a randomized clinical trial. NW PRECEDENT providers will invite subjects to participate if they are between the ages of 12 and 20 and have at least one new WSL on the 4 maxillary incisors associated with orthodontic treatment. These are the most common teeth to develop these lesions. The NW PRECEDENT provider must verify that the WSL were not present in the pre-orthodontic treatment records. Subjects must be willing to be placed into any of the following three groups:

1. Test Group A: 10% CPP-ACP + 900 ppm Fluoride paste - a trained staff member from the NW PRECEDENT dental/orthodontic office will give 3 tubes of MI Paste Plus and instructions to the subject for home use. The subjects will also receive non-prescription fluoride toothpaste (1100 ppm Fluoride) and oral hygiene instructions. The group will consist of 80 subjects, and each subject will be given enough MI Paste for the duration of the trial. Treatment will begin on the day of retainer delivery if the subject was recruited on the day of fixed appliance removal. Otherwise, the treatment will begin on the date of recruitment.
2. Test Group B: Fluoride Varnish Group - a trained staff member from the NW PRECEDENT dental/orthodontic office will provide a single fluoride varnish application (22,600 ppm Fluoride) to the subject. The subjects will also receive non-prescription fluoride toothpaste (1100 ppm Fluoride) and oral hygiene instructions. The group will consist of 80 subjects. Treatment will begin on the day of retainer delivery if the subject was recruited on the day of fixed appliance removal. Otherwise, the treatment will begin on the date of recruitment.
3. Control Group - These 80 subjects will receive non-prescription fluoride toothpaste (1100 ppm Fluoride) and oral hygiene instructions at the time of enrollment. After the trial is completed (~ August 2011), these subjects will be informed of the results, and offered one of the two active arms, if they are found to be effective in reducing WSL.

The NW PRECEDENT provider and the subject will also fill out a short survey to compile information about the subject's age, gender, race, ethnicity, time in fixed appliances, oral hygiene during treatment, and type of retainers after orthodontic treatment. Upon determining a subject's eligibility and willingness to participate, as well as obtaining assent/consent, he/she will be randomly assigned to a group, a baseline photograph will be taken, and the assigned treatment will begin. In the case of subjects who have just had their orthodontic appliances removed, the subjects will undergo enrollment and photos, but their assigned treatment will not begin until the day of retainer delivery. The subject's general dentist (if they did not perform their orthodontic care) will be sent a letter informing them that their patients are currently enrolled in the study, and that any additional treatment for white spot lesions should be delayed until the study is complete (8 weeks).

Subjects who are identified at some time after their fixed orthodontic appliances have been removed will have baseline photographs taken on the day of recruitment. Subjects who are identified on the day their appliances are removed will have photographs taken on that day, as well at the time of retainer delivery (2 - 7 days later). A subsequent analysis of the day of fixed appliance removal and one week follow-up photographs will be performed, in order to determine if significant changes are evident during this short period immediately after fixed appliance removal. This is being investigated because portions of the teeth under the braces have been shielded from the oral cavity for several years, and they may also have been desiccated during the removal of braces. Additionally, the gums may be puffy and swollen immediately after taking braces off, and parts of the teeth may not be visible. The photographs will be sent to the online data capture system.

At the eight-week time point, NW PRECEDENT providers will recall the subjects (240 total) and take the eight-week follow-up photographs in the same standardized format as the baseline photographs. The photographs will be sent via the online data capture system. The NW PRECEDENT provider will administer an in office survey to the subject to gather information regarding satisfaction with using the treatment, compliance, oral hygiene practices, and self-assessment of improvement of the WSL.

A group of blinded examiners consisting of five to ten laypersons and five to ten dental experts will view each subject's set of digital photographs in chronological order on a PowerPoint presentation. The photographs will only show the four maxillary incisor teeth and will be unidentifiable to the examiners. Each set of photographs will then be given an improvement rating on a 100 mm visual analog scale (VAS) (0=no improvement, 100=100% improvement). In addition, both a graduate orthodontic resident and a dental student will blindly assess the digital photographs by measuring the size of the white spot lesion relative to the rest of the tooth expressed as a percent. Statistical analysis will then be performed.

ELIGIBILITY:
Inclusion Criteria:

* Completed fixed appliance orthodontic therapy within the past two years
* Have at least one white spot lesion on the facial surface of a maxillary central or lateral incisor tooth that was not present prior to treatment with fixed orthodontic appliances.
* Between the ages of 12 and 20 years of age
* Agrees to randomization to the different treatment protocols
* Signed informed consent obtained from a parent or guardian of the patient f the patient is under the age of eighteen

Exclusion Criteria:

* Not willing to be randomly assigned to one of the three treatment groups
* Any abnormal oral, medical, or mental conditions, including any milk-related allergies and/or any medical conditions involving the kidneys.
* Any patients who underwent therapy for white spot lesion after completion of orthodontic treatment
* Any white spot lesion present on qualifying teeth with frank cavitation
* Patient is non-English speaking or non-English reading

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Improvement as rated by blinded assessors viewing photographs before and after treatment. | 8 weeks

SECONDARY OUTCOMES:
To investigate subjects' self-assessment of improvement against a group of blinded examiners for the amelioration of WSL. | 8 weeks
Improvement as rated by blinded assessors viewing photographs in the period between the day of orthodontic appliance removal and retainer delivery. | 2-7 days
To investigate variables (age, gender, time since fixed orthodontic appliance removal, compliance, oral hygiene practices, etc) that may influence WSL regression and the effectiveness of the treatment and control groups. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Greg H Huang, DMD,MSD,MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington/NW PRECEDENT, Seattle, Washington, United States